CLINICAL TRIAL: NCT04931953
Title: A Feasibility Trial of Neuromodulation With Connectivity-Guided Intermittent Theta Burst Stimulation for Cognitive Impairment in Multiple Sclerosis
Brief Title: Feasibility of Neuromodulation With Connectivity-Guided iTBS for Cognitive Impairment in MS
Acronym: TMS4MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21038
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be told whether they have been allocated to an active iTBS or sham iTBS administration until the end of their study participation, where they will be informed whether they received active or sham iTBS administration. The two technicians (including the research fellow) administering the iTBS will not be blind to group allocation.
  The RA conducting the cognitive assessments and analysing these (and the questionnaires) will be blinded to group allocation. We aim to stagger the commencement of the iTBS intervention schedule per group (with those in Group C [4-week intervention schedule] to begin first), to avoid participants returning for their EOI assessments 1, 2, or 4 weeks later depending upon group allocation. We hope that this will minimise the chance of unblinding the RA to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): iTBS intervention lasting 30 minutes, given 4 days a week, for 1 week
  Interventions: Other: Intermittent theta burst stimulation (iTBS)
- Group 2 (Active Comparator): iTBS intervention lasting 30 minutes, given 4 days a week, for 2 weeks
  Interventions: Other: Intermittent theta burst stimulation (iTBS)
- Group 3 (Active Comparator): iTBS intervention lasting 30 minutes, given 4 days a week, for 4 weeks
  Interventions: Other: Intermittent theta burst stimulation (iTBS)
- Group 4 (Sham Comparator): Sham iTBS intervention lasting 30 minutes, given 4 days a week, for 2 weeks.
  Interventions: Other: Sham Intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Other: Intermittent theta burst stimulation (iTBS) — The localisation of the left dorsolateral prefrontal cortex (DLPFC) target will be identified using effective connectivity of the left caudate to identify the maximally-connected locus in the left DLFPC. Following this the iTBS will be administered to the target coordinates identified using the neuronavigation software available with the system. Connectivity-guided iTBS is then administered using a 70mm Double Air Film Coil (Magstim, Whitland, Dyfed, UK), connected to a Magstim Super Rapid-2 Plus-1 stimulator. The administration comprises bursts of 3 pulses at 50Hz with a power of 80% motor threshold at a burst frequency of 5 Hz (i.e., every 200ms) for 2 seconds, repeated every 10 seconds for a total of 190 seconds (600 pulses). Blocks are repeated a total of 3 times, with 5-minute rest intervals between blocks. During left DLPFC stimulation, the TBS coil is held by a support tangentially to the skull, with the axis of the coil angled approximately 90 degrees from the midsagittal axis.
  Arms: Group 1; Group 2; Group 3
Other: Sham Intermittent theta burst stimulation (iTBS) — The sham iTBS administration is performed under the same conditions and with an identical protocol and equipment to the full administration, except that it uses a commercially available sham iTBS coil designed for use in double-blind trials. This sham coil looks like the real coil and connects to the iTBS unit but delivers only a very weak and shallow stimulation thus simulating the sounds made by the real iTBS coil.
  Arms: Group 4

SUMMARY:
Cognitive difficulties can affect many people who live with multiple sclerosis (MS). These difficulties, such as within thinking, memory, and problem solving, can have an impact on important aspects of an individual's life, including their daily activities, work, and how they manage their condition. Previous studies have suggested that cognitive difficulties affect approximately 40-70% of people living with MS, yet there are currently no treatments to target these problems. Recent research has directed towards a non-invasive intervention which stimulates a part of the brain (called the dorsolateral prefrontal cortex, or DLPFC for short) which is reported to participate in cognitive processes, such as memory, thinking, and attention. This intervention, called "intermittent theta burst stimulation" (iTBS), involves placing a magnetic device to the skull to activate the DLPFC underneath. This technique has been used successfully in the treatment of depression and is widely considered safe and painless. Previous studies have also shown that iTBS intervention can lead to improvements in cognitive processes.

Before the investigators can progress to a large trial to explore its clinical effectiveness for reducing cognitive problems for people with MS, some aspects regarding its feasibility need to be clarified, for example whether it is an acceptable and tolerable intervention for people living with MS. A single-centre, mixed methods feasibility randomised controlled trial will be conducted to compare four groups (10 participants each) of iTBS administration. At baseline, End of Intervention (EOI), and 8-week follow up, the investigators will complete outcome measures to evaluate cognition, mood and fatigue. Participants will also undergo MRI scans at baseline and EOI. Following participation, participants will be interviews and the investigators will organise a post-participation workshop to explore their experiences of the trial, including the tolerability of the protocol and acceptability of the visit schedule, and any differences in cognition.

DETAILED DESCRIPTION:
The primary objective is to assess the feasibility of the trial procedures, in terms of their acceptability and tolerability for pwMS who have cognitive impairment. For this aim, the completion of the intervention schedule will be measured (e.g., attending all sessions per the protocol, considering any missed appointments and reasons for non-attendance where possible) including the end of intervention assessments, as well as the 8-week follow up to ascertain participant willingness to complete the full study.

Participants will be randomly allocated to one of four groups (Group 1: 4 administrations of intermittent theta burst stimulation (iTBS) over 1 week; Group 2: 8 administrations of iTBS over 2 weeks; Group 3: 16 administrations of iTBS over 4 weeks; Group 4: 8 administrations of sham iTBS over 2 weeks). Participants will not be aware whether they have been allocated to receive active or sham iTBS administration.

Intervention - Active iTBS: Active connectivity-guided iTBS will be administered to the left dorsolateral prefrontal cortex (DLPFC). The administration comprises bursts of 3 pulses at 50Hz with a power of 80% motor threshold, at a burst frequency of 5 Hz (i.e., every 200ms) for 2 seconds, repeated every 10 seconds for a total of 190 seconds (600 pulses). Blocks are repeated a total of 3 times, with 5 minutes rest intervals between blocks. (Duration and frequency: 30 min, 4 times a week for up to 4 weeks depending on group).

Sham iTBS: The sham iTBS administration is performed under the same conditions and with an identical protocol and equipment to the full administration, except that it uses a commercially available sham iTBS coil designed for use in double-blind trials. This sham coil looks like the real coil and connects to the iTBS unit but delivers only a very weak and shallow stimulation thus simulating the sounds made by the real iTBS coil.

At baseline, End of Intervention (EOI), and 8-week follow up, outcome measures will be completed to evaluate cognition, mood and fatigue. Participants will also undergo MRI scans at baseline and EOI. The purpose of the MRI is to allow identification of the exact location over which the iTBS intervention will be applied, and it will allow measurement of brain function before iTBS intervention (or sham).

The MRI scan will include:

* High resolution T1-weighted structural brain image for image co-registration,
* Resting-state functional MRI (rs-fMRI) for connectivity-guided neuronavigation,
* Fluid attenuated inversion recovery (FLAIR)
* Diffusion tensor imaging (DTI) acquisitions to quantification spatial mapping of macro- and mircrostructural white matter injury,
* Arterial Spin Labelling (ASL) perfusion imaging to map cerebral blood flow.
* Task related functional MRI - N-Back task.

The investigators have developed a questionnaire to explore tolerability and acceptability of the procedures, and participants will also be invited to discuss their experience of participating in the trial at interview 8 weeks post-intervention.

Finally, at the end of the study, the investigators aim to host a post-participation workshop at the beginning of month 28, following collection and analysis of main outcomes. Depending on covid-safe recommendations from the government and university, this may be via video call or at a venue. All participants will be invited to discuss whether the experience of participation (varying from 1-week to 4-weeks) can inform which of intervention regime investigators should take forward into a subsequent pilot trial, to expand on the preliminary data analysis from the qualitative interviews. Investigators will explore the magnitude and nature of the effect on cognition that would be needed to be achieved to give a meaningful change to them personally, such that the iTBS interventions of different durations would be warranted. For example, participants may feel that only a major improvement in day-to-day cognition would justify a 4-week intervention, whereas others may feel that any benefit would justify this. These issues will be explored to inform future trial design.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 - 69 years.
* Received a diagnosis of MS (any type of MS) at least 12 months prior to baseline assessment.
* Report cognitive problems, as determined by a cut-off score of 55 or lower on the oral SDMT
* Ability to give informed consent
* Able to commit to regular attendance in clinic, for up to 4 times a week for 4 weeks and follow up appointment eight weeks after the end of trial procedures.

Exclusion Criteria:

* Diagnosed with depression or scores ≥15 on the Patient Health Questionnaire-9
* Medical history of, or self-reported, seizures
* Neurological conditions (in addition to MS), e.g., brain neoplasm, cerebrovascular events, epilepsy, prior brain injury or brain surgery
* Contraindications to MRI scanning (identified by standard MRI safety screening questionnaire).
* Contraindications to TMS, including hairstyles or piercings that would impair magnetic transmission which cannot be altered to ensure effective intervention
* Frequent panic attacks which are likely to prevent regular attendance or participation in MRI/TMS procedures
* Prior TMS intervention
* Pregnancy
* MS relapse within the preceding 6 weeks
* Significant mobility problems if they are likely to preclude regular attendance in clinic, for up to 4 times a week for 4 weeks
* Involved with any other clinical trials involving medical procedures, interventions or treatment.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Trial Procedures | 8 weeks
  Number of sessions attended according to the protocol Number of missed/rescheduled appointments Reasons for non-attendance Completion of end of intervention assessments Completion of 8 weeks follow up assessments

SECONDARY OUTCOMES:
Feasibility of recruitment | 1 week
  Proportion of eligible and consenting participants
The Brief Visuospatial Memory Test Revised (BVMT-R) Trials 1-3. | 8 weeks
  Raw scores range from 0 to 12 for each trial and reflect accuracy and correct placement (higher scores indicate better outcome)
The Brief Visuospatial Memory Test Revised (BVMT-R) Total learning | 8 weeks
  Sum of scores across the three trials (min: 0, max: 36; higher scores indicate better outcome).
The Brief Visuospatial Memory Test Revised (BVMT-R) Learning | 8 weeks
  The best of Trial 2 or 3 minus the Trial 1 score (min 0 max 23, higher scores indicate better outcome)
The Brief Visuospatial Memory Test Revised (BVMT-R) Delayed recall | 8 weeks
  Raw scores range from 0 to 12 (max) and reflect recall of designs after 25-min delay. Higher scores indicate better outcome.
The Brief Visuospatial Memory Test Revised (BVMT-R) Percent retained | 8 weeks
  Scores range from 1 to 100 (max) and reflect the amount originally learned that was retained across the delay. Higher scores indicate better outcome.
The Brief Visuospatial Memory Test Revised (BVMT-R) Recognition hits | 8 weeks
  - Number of target figures correctly recognized; scores range from 0 to 6 (max). Higher scores indicate better outcome.
The Brief Visuospatial Memory Test Revised (BVMT-R) Recognition false alarms | 8 weeks
  Number of distractors incorrectly recognized as targets; scores range from 0 to 6 (max). Higher scores indicate better outcome.
The Brief Visuospatial Memory Test Revised (BVMT-R) Recognition discrimination index | 8 weeks
  Recognition hits minus recognition false alarms; scores range from -6 to 6 (max). Higher scores indicate better outcome.
The Brief Visuospatial Memory Test Revised (BVMT-R) Recognition response bias | 8 weeks
  Scores range from 0.00 to 1.00 (max) and reflect the tendency (or lack of) to answer "yes" to a recognition item. Higher scores indicate better outcome.
The California Verbal Learning Test-II (CVLT-II) | 8 weeks
  A computer administration and scoring system generates score, graphs a learning curve, and provides learning parameters, response errors and interference effects. Higher scores indicate better outcome.
The Symbol Digit Modalities Test (SDMT) | 8 weeks
  Raw score of correct items named per 90 seconds. Minimum value: 0 Maximum value: 130. Higher scores indicate better outcome.
Digit Span Forwards (from WAIS-IV) | 8 weeks
  Raw score, minimum 0, maximum 16. Higher scores indicate better outcome.
Digit Span Backwards (from WAIS-IV) | 8 weeks
  Raw score, minimum 0, maximum 16. Higher scores indicate better outcome.
Patient Health Questionnaire - Depression | 8 weeks
  Self-rated mood. Raw score, minimum 0, maximum 27. Lower scores indicate better outcome.
General Anxiety Disorder Scale | 8 weeks
  Self-rated anxiety. Raw score, minimum 0, maximum 21. Lower scores indicate better outcome.
Perceived Deficits Questionnaire (PDQ) | 8 weeks
  Self-reported cognitive impairment. Raw score, minimum 0, maximum 80. Lower scores indicate better outcome.
The Modified Fatigue Impact Scale (MFIS) | 8 weeks
  Self-reported fatigue. Raw score, minimum 0, maximum 84. Lower scores indicate better outcome.
The Edinburgh Handedness Inventory (EHI) | 1 week
  Self-rated handedness to determine whether one favours left or right-handedness. It is not scored; result will be binary (left/right).
Change in effective connectivity between left dorsolateral prefrontal cortex and left caudate nucleus | 5 weeks
  As above
Change in cerebral blood flow in the left dorsolateral prefrontal cortex and in the left caudate nucleus (normalised to whole brain cerebral blood flow) | 5 weeks
  As above
Safety outcomes of iTBS | 4 weeks
  Number of participants with treatment-related adverse events and number of events each, as reported to research team
Undesired effects of iTBS | 4 weeks
  Number of participants with self reported negative effects e.g., headaches, dizziness
iTBS Experience Questionnaire - Tolerability | 1 week
  Unpleasant sensations of iTBS. Minimum score 0, maximum score 15. Higher indicates worse outcome.
iTBS Experience Questionnaire - Acceptability | 1 week
  Minimum score 0, maximum score 30. Higher score indicates better outcome.
iTBS Experience Questionnaire - Blinding | 1 week
  Number of participants who correctly guessed allocation to sham/active iTBS intervention
Interviews - Tolerability | 1 week
  Tolerability of the trial procedures - qualitative analysis via framework method
Interviews - Acceptability | 1 week
  Acceptability of the trial procedures of the trial procedures- qualitative analysis via framework method
Interviews - perceived differences | 1 week
  Subjective perceived differences in cognitive abilities in daily life - qualitative analysis via framework method
Interviews - Improvements | 1 week
  Suggested improvements to refine trial procedures - qualitative analysis via framework method
Post-participation workshop | 1 week
  A semi-structured focus group schedule will explore qualitative data regarding meaningful changes to cognition/mood and how much change would be expected given the requirements of the intervention at the post-participation workshop. This will be analysed using framework analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided